CLINICAL TRIAL: NCT06340113
Title: Comparison of Mulligan and McKenzie Exercises Along With Stabilization Exercises on Pain, Range of Motion and Disability in Patients With Chronic Neck Pain
Brief Title: Mulligan and Mckenzie Exercises Alongwith Stabilization Exercises in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0108 NASHIA
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
Keywords: Disability, Mulligan mobilizations, Neck pain, Pain
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCKENZIE AND STABILIZATION EXERCISES (Experimental): In this group, 11 participants will be included. the interventions will be given for 15 mint. The exercises then repeated five or six times in a Session. the session will be of 45 mins, 3 session per week
  Interventions: Procedure: MCKENZIE AND STABILIZATION EXERCISES
- MULLIGAN AND STABILIZATION EXERCISES (Experimental): In this group, 11 participants will be included. the interventions will be given for 15 mint. The exercises then repeated five or six times in a Session. the session will be of 45 mins, 3 session per week for 10 weeks
  Interventions: Procedure: MULLIGAN AND STABILIZATION EXERCISES

INTERVENTIONS:
Procedure: MCKENZIE AND STABILIZATION EXERCISES — In this group 11 participants will receive McKenzie protocol with stabilization exercises. Participants will be asked to sit to treat extension deficit. The participant will be in a comfortable sitting position with a proper back support. Head is kept in forward facing without any up and done movement (10 to 15 times). Then, he restored the neutral sitting posture, and at the end of the range of motion (ROM), he' tuck in" chin by pushing the chin with his fingers (10 to 15 times). The exercises then repeated five or six times in a Session. the session will be of 45 mins, 3 session per week. At end of each session patients will do stabilization exercises with 10reps of each exercise with 10sec hold
  Other Names: MCKENZIE PROTOCOL AND RHYTHMICAL STABILIZATION EXERCISES
  Arms: MCKENZIE AND STABILIZATION EXERCISES
Procedure: MULLIGAN AND STABILIZATION EXERCISES — . The technique will include Self-sustained Natural Apophyseal Glide (SNAGs), Natural Apophyseal Glides (NAGs), and mobilization techniques.. The participants will receive three sets of Mulligan Mobilization, each set involving 10 repetitions of the exercise, with an interval of 15 to 20 seconds between the sets.At end of each session patients will do stabilization exercises with 10reps of each exercise with 10sec hold.
  Other Names: MULLIGAN AND RHYTHMICAL STABILIZATION EXERCISES
  Arms: MULLIGAN AND STABILIZATION EXERCISES

SUMMARY:
The goal of this [type of study: Randomized control trial] is to [ compare the effectiveness of Mulligan and McKenzie Exercises along with stabilization exercises on pain, range of motion and disability ] in [ in patients with chronic neck pain].The main question it aims to answer is:

* Wether Mulligan is more effective or Mckenzie exercises along with stabilization exercises in the treatment of patients with chronic neck pain Group 1 will recieve Mulligan and stabilization exercises Group 2 will recieve Mckenzie and stabilization exercises

DETAILED DESCRIPTION:
Chronic neck pain is a prevalent and multifaceted condition, affecting a substantial portion of the general population (16.7% to 75.1%). Different techniques have been used to treat chronic neck pain. In this study, I will be comparing two manual therapy techniques along with stabilization exercises and will check which manual technique with stabilization exercise is more effective in the treatment of chronic neck pain. One of the techniques is Mulligan technique. The other one is the self-treatment approach of the McKenzie technique, . Additionally, cervical stabilization exercises, incorporating progressive stages, aim to enhance neuromuscular control.

The research involves two intervention groups (Group A and Group B) receiving specific treatments over 32 sessions within an eight-week period. Group A incorporates the Mulligan technique, cervical and scapulothoracic stabilization exercises, and transcutaneous electrical nerve stimulation (TENS) with a heating pad. Group B undergoes hot packs and TENS, followed by McKenzie exercises and cervical and scapulothoracic stabilization exercises. Outcomes, encompassing pain levels, range of motion (ROM), and Neck Disability Index (NDI) scores, will be evaluated using the Numeric Pain Rating Scale, Goniometer, and Neck Disability Scale. Data analysis will employ SPSS version 26. Data will be collected at baseline, immediately post-intervention, and at follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 Localized chronic neck pain for more than 3 months

Exclusion Criteria:

* Participants suffering their neck pain was caused by any other complications.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4weeks
  NPRS consists of a scale with 0-10 readings. The zero denotes no pain while 1, 2, 3 denotes to mild pain, 4, 5, 6 denotes to moderate pain while 7-10 denotes to severe pain.
Neck Disability Index (NDI) | 4 WEEKS
  The NDI consists of ten questions. Each question has six different assertions expressing progressive levels of pain or limitation in activities. Item scores range from 0 (no pain or limitation) to 5 (as much pain as possible or maximal limitation). The total NDI score ranges from 0 to 5 points. Higher scores indicate greater disability.
Goniometer | 4 weeks
  Active Range of Motion of the patient will be assessed using a universal standard goniometer for cervical flexion, extension, side flexion (left and right), rotation (left and right). The data will be collected at baseline cervical goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, ms, Principal Investigator — riphah lahore
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No